CLINICAL TRIAL: NCT00000846
Title: A Phase I Trial To Evaluate the Safety and Immunogenicity of the UBI HIV-1MN PND Peptide Immunogen, Given by IM Injection, in Combination With the UBI Microparticulate Monovalent HIV-1 MN Branched Peptide Given Orally, in HIV-1 Uninfected Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 023
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV-1; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: HIV-1 Peptide Vaccine, Microparticulate Monovalent
Biological: HIV-1 Peptide Immunogen, Multivalent

SUMMARY:
To evaluate safety and immunogenicity of 2 different HIV-1 peptide candidate vaccines, the UBI HIV-1 MN PND peptide immunogen and the UBI microparticulate monovalent HIV-1 MN branched peptide when administered sequentially by 2 different routes of immunization, parental priming followed by oral boosting.

DETAILED DESCRIPTION:
After the prescreening, volunteers will be randomized into Group I or Group II. Each group will contain 16 volunteers. At least 5 volunteers in each group must be women. At month 0 all volunteers will receive multivalent HIV-1 peptide immunogen or the placebo. Group I will receive the injection in the deltoid and Group II will receive it in the anterior thigh. At months 1, 2 and 8 all patients will receive microparticulate monovalent HIV-1 peptide or the placebo. Follow up will be conducted.

ELIGIBILITY:
Inclusion Criteria

Patients must have or be:

* Healthy.
* Negative ELISA for HIV.
* Negative for Hepatitis B surface antigen.
* Normal urine dipstick.
* Normal history and physical exam.
* Availability for follow-up for planned duration of the study (60 weeks).

Risk Behavior: Required:

* Lower or intermediate risk sexual behavior as defined by AVEG.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Medical or psychiatric condition or occupational responsibilities which preclude subject compliance with the protocol.
* Active syphilis. NOTE: If the serology is documented to be a false positive or due to a remote (> 6 months) treated infection, the volunteer is eligible.
* Active tuberculosis. NOTE: Volunteers with a positive PPD and a normal chest X-ray showing no evidence of TB and not requiring INH therapy are eligible.

Patients with any of the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, malignancy or autoimmune disease.
* History of anaphylaxis or other serious adverse reactions to vaccines.
* History of inflammatory gastrointestinal disease, celiac disease or intestinal malignancy.
* History of acute gastroenteritis within the past month or gastrointestinal surgery within the past 12 months.

Prior Medication:

Excluded:

* History of use of immunosuppressive medication.
* Live attenuated vaccines within 60 days of study. NOTE: Medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) are not exclusionary but should be given at least 2 weeks away from HIV immunizations.
* Use of experimental agents within 30 days prior to study.
* Receipt of blood products or immunoglobulin in the past 6 months.
* Prior receipt of HIV vaccines or a placebo recipient in an HIV vaccine trial.

Risk Behavior:

Excluded:

* Subjects with identifiable higher risk behavior for HIV infection as determined by screening questionnaire designed to identify risk factors for HIV infection.
* History of injection drug use within the last 12 months to enrollment.
* Higher risk sexual behavior as defined by AVEG.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36

CONTACTS AND LOCATIONS:
Overall Officials: Mulligan M, Study Chair
Locations (3):
- United States (3):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Rochester Med Ctr, Rochester, New York
  - Univ of Washington / Pacific Med Ctr, Seattle, Washington